CLINICAL TRIAL: NCT04659928
Title: Evaluation of Aerosol in a Dental Clinic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Claudia Ruiz Brisuela, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-DB-20-1017
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- High volume evacuation (HVE) suction only and hydrogen peroxide (Experimental)
  Interventions: Device: High volume evacuation (HVE); Drug: Hydrogen Peroxide
- HVE suction and extraoral vacuum aspirator (EVA) and hydrogen peroxide (Experimental)
  Interventions: Device: High volume evacuation (HVE); Device: Extraoral vacuum aspirator (EVA); Drug: Hydrogen Peroxide
- HVE suction and extraoral vacuum aspirator (EVA) and Placebo (Experimental)
  Interventions: Device: High volume evacuation (HVE); Device: Extraoral vacuum aspirator (EVA); Drug: Placebo
- High volume evacuation (HVE) suction only and Placebo (Experimental)
  Interventions: Device: High volume evacuation (HVE); Drug: Placebo

INTERVENTIONS:
Device: High volume evacuation (HVE) — Intra oral suction will be done and during the procedure,bacterial colony forming units (cfus) will be captured during dental care by placing large format petri dishes containing bacterial culture media in the dental operatory with open lids. Once aerosol capture is complete, petri dishes will be incubated and quantified under BSL-2 safety conditions in the lab. Patient will be given a mouth rinse.
Device: Extraoral vacuum aspirator (EVA) — Extraoral suction connected to dental suction will be used and bacterial colony forming units (cfus) will be captured during dental care by placing large format petri dishes containing bacterial culture media in the dental operatory with open lids. Once aerosol capture is complete, petri dishes will be incubated and quantified under BSL-2 safety conditions in the lab. Patient will be given mouth rinse.
  Arms: HVE suction and extraoral vacuum aspirator (EVA) and Placebo; HVE suction and extraoral vacuum aspirator (EVA) and hydrogen peroxide
Drug: Hydrogen Peroxide — Subjects will be given 1.5 % Oral Solution of hydrogen peroxide mouth rinse
  Arms: HVE suction and extraoral vacuum aspirator (EVA) and hydrogen peroxide; High volume evacuation (HVE) suction only and hydrogen peroxide
Drug: Placebo — Subjects will be given a placebo (plain water) mouth rinse
  Arms: HVE suction and extraoral vacuum aspirator (EVA) and Placebo; High volume evacuation (HVE) suction only and Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of external evacuation units and mouth rinses during aerosol generating procedures in a dental clinic and to determine the risk level to the dental practitioners during aerosol generating procedures.

ELIGIBILITY:
Inclusion Criteria:

* prepping natural teeth at the appointment
* at least an hour long procedure
* procedure will be the first one in the morning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ruiz Brisuela, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
Started | 10 | 10 | 11 | 10
Completed | 10 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo | Total
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 7 | 9 | 26
  >=65 years | 6 | 4 | 4 | 1 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 5 | 17
  Male | 7 | 6 | 6 | 5 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Bacterial Colony Forming Units (CFUs)
Description: At baseline (1 hour before treatment), four agar petri dishes will be placed at standardized distances (2 ft, 3 ft, 4 ft, and 6 ft) from the dental chair headrest in the operating room. An impinger will also be positioned 2 ft from the headrest. The number of bacterial colony-forming units (CFUs) will be counted for each petri dish and the impinger after a 72-hour incubation period. The average number of Bacterial CFUs is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: bacterial colony forming units (CFUs)
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
Number analyzed (Participants) | 10 | 10 | 11 | 10
bacterial colony forming units (CFUs) | 47.2 (16.38) | 125.3 (155.43) | 70.7 (98.06) | 116.7 (143.38)

2. Secondary Outcome: Number of Bacterial Colony Forming Units (CFUs) at Each Location
Description: At baseline (1 hour before treatment), four agar petri dishes will be placed at standardized distances (2 ft, 3 ft, 4 ft, and 6 ft) from the dental chair headrest in the operating room. An impinger will also be positioned 2 ft from the headrest. The number of bacterial colony-forming units (CFUs) will be counted for each petri dish and the impinger after a 72-hour incubation period. The number of Bacterial CFUs per location is reported
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Bacterial Colony Forming Units (CFUs)
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
Number analyzed (Participants) | 10 | 10 | 11 | 10
Bacterial Colony Forming Units (CFUs)
  Impinger (2 feet from dental chair headrest) | 0.6 (0.96) | 33.4 (93.86) | 2.22 (3.34) | 35.11 (99.36)
  Plate 1 (2 feet from dental chair headrest) | 13 (8.51) | 10.8 (8.53) | 9.22 (5.38) | 18.44 (30.61)
  Plate 2 (3 feet from dental chair headrest) | 12.3 (9.63) | 7.3 (5.51) | 40.66 (97.39) | 11.11 (5.27)
  Plate 3 (4 feet from dental chair headrest) | 10.7 (6.37) | 66.2 (123.33) | 9 (6.72) | 11.66 (14.80)
  Plate 4 (6 feet from dental chair headrest) | 10.6 (7.84) | 7.6 (6.07) | 9.66 (6.63) | 40.44 (97.47)

3. Secondary Outcome: Number of Bacterial Colony Forming Units (CFUs) at Each Location
Description: At the start of treatment, four agar petri dishes will be placed at standardized distances (2 ft, 3 ft, 4 ft, and 6 ft) from the dental chair headrest in the operating room for one hour. An impinger will also be positioned 2 ft from the headrest for one hour. The number of bacterial colony-forming units (CFUs) will be counted for each petri dish and the impinger after a 72-hour incubation period. The number of Bacterial CFUs per location is reported.
Time Frame: 1 hour from the start of the treatment
Measure: Mean (Standard Deviation); unit: Bacterial Colony Forming Units (CFUs)
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
Number analyzed (Participants) | 10 | 10 | 11 | 10
Bacterial Colony Forming Units (CFUs)
  Impinger (2 feet from dental chair headrest) | 31.4 (94.39) | 31.3 (94.43) | 2.9 (3.34) | 3.44 (5.36)
  Plate 1 (2 feet from dental chair headrest) | 9.4 (4.50) | 16.9 (28.33) | 11.5 (6.98) | 12.33 (7.46)
  Plate 2 (3 feet from dental chair headrest) | 10.8 (8.10) | 14.5 (16.09) | 13.2 (11.28) | 12.11 (9.58)
  Plate 3 (4 feet from dental chair headrest) | 40.3 (91.59) | 11.3 (8.05) | 10.2 (3.11) | 12.22 (8.54)
  Plate 4 (6 feet from dental chair headrest) | 9.4 (5.31) | 13.1 (12.99) | 7.9 (6.06) | 12.33 (8.42)

4. Primary Outcome: Number of Bacterial Colony Forming Units (CFUs)
Description: At the start of treatment, four agar petri dishes will be placed at standardized distances (2 ft, 3 ft, 4 ft, and 6 ft) from the dental chair headrest in the operating room for one hour. An impinger will also be positioned 2 ft from the headrest for one hour. The number of bacterial colony-forming units (CFUs) will be counted for each petri dish and the impinger after a 72-hour incubation period. The average number of Bacterial CFUs is reported.
Time Frame: 1 hour from the start of the treatment
Measure: Mean (Standard Deviation); unit: bacterial colony forming units (CFUs)
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
Number analyzed (Participants) | 10 | 10 | 11 | 10
bacterial colony forming units (CFUs) | 101.3 (131.9) | 87.1 (101) | 45.7 (15.28) | 52.44 (17.89)

ADVERSE EVENTS:
Time Frame: Up to 1 hour
Arm/Group | High Volume Evacuation (HVE) Suction Only and Hydrogen Peroxide | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Hydrogen Peroxide | High Volume Evacuation (HVE) Suction Only and Placebo | HVE Suction and Extraoral Vacuum Aspirator (EVA) and Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT04659928/Prot_SAP_000.pdf